CLINICAL TRIAL: NCT04478240
Title: Automating Peer Learning to Reduce Alcohol Use and Related Deviant Behavior in Secondary School
Acronym: PeerLearning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AA027422
Record Dates: First submitted 2020-07-06; First posted 2020-07-20 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Substance Use; Stress; Relation, Interpersonal; Bullying; Victimisation; Mental Health Issue; Sleep, Inadequate; Social Skills
Keywords: Cooperative learning; Deviant peer affiliation; School-based prevention; Alcohol and other drug use; Adolescence Middle/high school; Mental health; Stress; Sleep quality; Bullying; Victimization; Social-Emotional Learning (SEL); Educational technology
MeSH Terms: conditions — Substance-Related Disorders; Bullying; Sleep Deprivation; Social Skills; Psychological Well-Being; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized trial, where assignment to condition occurs at the school level. Randomization of schools to condition (intervention vs. control) occurs at the beginning of the study and there is no cross-over.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (access to PeerLearning.net) (Experimental): Teachers and students in intervention schools will be given access to PeerLearning.net software for the purposes of instruction for the 2021-2022 school year.
  Interventions: Behavioral: PeerLearning.net
- Passive Control (no intervention) (No Intervention): Teachers and students in control schools will conduct instruction as usual without PeerLearning.net.

INTERVENTIONS:
Behavioral: PeerLearning.net — PeerLearning.net is a software package that supports teachers in designing and delivering peer learning lessons, either in-person or remotely while students are learning at home.
  Peer learning is an instructional technique that puts students in groups under conditions of positive interdependence, where they are incentivized to work together and promote the success of one another. Peer Learning lessons also ensure individual accountability and explicitly observe for and reward specific group social skills (e.g., encouraging participation, checking for understanding). Peer Learning also includes group processing after the lesson is completed so that the students in the groups have an opportunity to discuss what they did well and what could use improvement; they also have the opportunity to provide positive reinforcement to one another for contributing to the success of the group.
  Arms: Intervention (access to PeerLearning.net)

SUMMARY:
Deviant peer affiliation is one of the most important predictors of alcohol use in adolescence. These affiliations arise when socially marginalized youth self-aggregate and reinforce alcohol use and other deviant activity (i.e., "deviant peer clustering"). Existing efficacious school-based prevention programs generally have small effects and can be difficult to disseminate with fidelity and challenging to sustain due to complex designs and significant time-and-money expenditures required for materials and training. Existing school-based prevention programs have not provided compelling value to schools, which has limited their dissemination. The investigators found significantly lower rates of deviant peer affiliation and alcohol/tobacco use and moderate-to-strong suppressive effects on bullying, victimization, stress, and emotional problems, and strong positive effects on student engagement, achievement, and social-emotional skills in peer-learning intervention schools compared to control schools. However, teachers in intervention schools faced challenges implementing peer learning, including: (1) design fidelity: ensuring that peer learning provided the most positive student experience by including all the essential design elements; and, (2) instructional support: managing the flow and timing of the activities to complete the lesson on time while dealing with unexpected disruptions. Investigators developed an initial version of a mobile software application (PeerLearning.net) that provided easy-to-use organizational templates with workflow support that teachers used to automate the design and delivery of peer learning lessons. In this cluster randomized trial of the app, the investigators will use a sample of middle and high schools and conduct pre/post student assessments of peer relations, alcohol/drug use, antisocial/prosocial behavior, and social-emotional skills. They will also collect information on stress, bullying/victimization and related outcomes, including sleep quality and mental health. Investigators will also collect data on the frequency of lesson delivery with the app by teacher and school to assess dosage, which will be incorporated into our analyses. The investigators hypothesize that use of PeerLearning.net will have significant suppressive effects on alcohol use and related outcomes (i.e., tobacco/marijuana use, antisocial behavior, bullying, emotional problems) and promote increased levels of social-emotional skills and prosocial behavior. The investigators hypothesize that these results will be moderated by dosage (i.e., use of the app), such that greater usage yields larger effects.

DETAILED DESCRIPTION:
Schools (N = 12) will be randomly assigned to intervention or waitlist control conditions, and data will be collected immediately in the fall (i.e., baseline measure) and in the spring, approximately 6 months later (i.e., post-treatment assessment). Overall, the investigators will have two assessment points. Data will be collected from teachers and students via on-line surveys (i.e., Qualtrics) and through observations; see below on the Measures. Intervention schools will receive training and access to the PeerLearning.net app immediately, whereas control schools will receive access in the spring after the second wave of data collection is completed.

The investigators hypothesize that usage of PeerLearning.net will promote increasing levels of prosocial behavior and have a significant suppressive effects on alcohol use and related outcomes (i.e., tobacco/marijuana use, antisocial behavior, bullying/victimization, mental health problems) and salutary effects on social-emotional skills, peer relations, and sleep quality. The investigators hypothesize that there will be effects of dosage (i.e., usage of the app). Finally, the investigators will examine differences in program effects by sex (gender) and ethnicity, which the investigators expect to be small or nonexistent.

Participants will include both teachers and students at 12 middle and high schools, cluster randomized to intervention vs. waitlist control. Teachers will use PeerLearning.net to design and deliver small-group peer learning lessons during the school year. The investigators will not exclude any participant based upon race/ethnicity, gender, or disability. Participating schools, teachers, and students will be rewarded.

ELIGIBILITY:
Inclusion Criteria:

* All teachers and students in participating schools will be eligible to participate.

Exclusion Criteria:

* The investigators will not exclude any participant based upon race/ethnicity, gender, or disability.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 924 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Alcohol and other drug (AOD) use | Pre and 6 months post-treatment
  Youth will complete the SAMHSA Participant Outcome Measures for Discretionary Programs. This survey tool was used as part of SAMHSA's national cross-site evaluation and is comprised of questions that include alcohol, tobacco, and other drug (ATOD) use and knowledge; ATOD beliefs and perceived risk of harm from ATOD use; and future intentions to use drugs. The investigators will also assess binge alcohol use (i.e., occasions at which 5/more drinks were consumed). The minimum score is zero.
Antisocial/prosocial behavior and mental health | Pre and 6 months post-treatment
  The Strengths and Difficulties Questionnaire (SDQ),has subscales for Conduct Problems (antisocial behavior), Prosocial Behavior, and Emotional Problems. Subscales for conduct problems (e.g., "I get very angry and often lose my temper"), emotional problems (e.g., "I worry a lot"), and prosocial behavior (e.g., "I usually share with others") items scores 1 (none) to 3 (a lot), and the investigators average these, so the minimum is 1 and the maximum is 3.
Bullying and victimization | Pre and 6 months post-treatment
  The Illinois Aggression Scales (Espelage & Holt, 2001) includes three subscales. The bullying and victimization subscales will be used. The 9-item Illinois Bully Scale measures frequency of teasing, name-calling, and social exclusion within the last 30 days. The 4-item Illinois Peer Victimization Scale assesses verbal and physical peer victimization within the past 30 days. Each item scores between 0 (none) and 4 (a lot), and the investigators average these so the minimum score is zero and the maximum is 4.
Sleep quality | Pre and 6 months post-treatment
  Pittsburgh Sleep Quality Inventory (PSQI) contains a series of items for sleep duration, sleep onset latency, and perceived sleep quality. Higher scores indicate greater duration, latency, and quality.
Stress | Pre and 6 months post-treatment
  Perceived Stress Scale (PSS); items are scored from 1 to 4 and averaged. Higher scores indicate more stress.
Peer support | Pre and 6 months post-treatment
  Classroom Life Scale; items are scored from 1 to 5 and averaged. Higher scores indicate more peer support.
Peer relations | Pre and 6 months post-treatment
  Peer Relatedness Scale items are scored from 1 to 4 and averaged. Higher scores indicate more positive peer relations.
Social-emotional skills | Pre and 6 months post-treatment
  Social and Emotional Competency Long-Form Assessment contains five subscales corresponding to the 5 dimensions of Social-Emotional Learning (Self-Awareness: a person's ability to recognize their emotions, thoughts, and values; Self-Management: a person's ability to regulate their emotions, thoughts, and behaviors; Social Awareness: the ability to recognize and empathize with others' perspectives and understand social norms; Relationship Skills: the ability to communicate and cooperate effectively, and to seek and offer help when needed; and Responsible Decision-Making: the ability to make constructive personal choices in relation to social norms and personal safety). Items are scored from 1 to 4 and averaged, with higher scores indicating greater social-emotional skill.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Espelage DL, Holt MK. Bullying and Victimization During Early Adolescence, Journal of Emotional Abuse. 2001. 2:2-3, 123-142, DOI: 10.1300/J135v02n02_08
- [Derived] Chirimwami V, Van Ryzin MJ. Universal School-Based Substance Use Prevention Using Technology-Supported Cooperative Learning. Prev Sci. 2024 Apr;25(3):488-497. doi: 10.1007/s11121-024-01662-1. Epub 2024 Mar 1. PMID 38427269